CLINICAL TRIAL: NCT05867966
Title: Evolution and Management of a Psychoneurological Symptom Cluster in Patients Who Had a Breast Cancer or a Digestive Cancer
Brief Title: Psychoneurological Symptom Cluster in Oncology
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Liege (Other)
Collaborators: Centre Hospitalier Universitaire de Liege (Other); Fonds pour la Recherche Scientifique (FRS-FNRS) (Unknown)
Responsible Party: Principal Investigator, Audrey Vanhaudenhuyse, PhD, University of Liege
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PNSC_onco
Record Dates: First submitted 2023-04-27; First posted 2023-05-22 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Cancer; Breast Cancer; Digestive Cancer
Keywords: cancer; oncology; symptoms; quality of life; hypnosis; self-care
MeSH Terms: conditions — Neoplasms; Breast Neoplasms; Gastrointestinal Neoplasms

STUDY DESIGN:
Intervention Model Description: The WP1 is observational only (N = 440) In the WP2, 60 other participants will be randomized into an intervention group and a control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): These participants will benefit from an 8-week group intervention combining psychoeducation, self-care learning and hypnosis exercises.
  Interventions: Behavioral: psychoeduc/self-care/self-hypnosis group
- Control group (No Intervention): These participants will not benefit from any intervention. After the end of the study, they will have the possibility to participate in the group intervention if they want to.

INTERVENTIONS:
Behavioral: psychoeduc/self-care/self-hypnosis group — See arm description.
  Arms: Intervention group

SUMMARY:
A psychoneurological symptom cluster is increasingly documented in oncology. It is composed of cancer-related fatigue, sleep difficulties, pain, emotional distress, and cognitive difficulties. These symptoms are linked by strong but complex relationships, and reinforce each other, negatively impacting patients' quality of life and survival. The configuration of this cluster (i.e., the relationships between the symptoms) seems different according to the cancer diagnosis or moment in the cancer journey. It has however been very little studied. Network analysis is an innovative method that allows a deeper understanding of the interactions between these symptoms. It also allows to compare patterns of clustering between distinct populations or measurement times. Finally, it allows to determine one core symptom in a cluster (i.e., the one with the strongest associations with the other symptoms), which could represent a target of choice for interventions aiming to improve the whole symptom cluster. This innovative project has then two main goals. First, the investigators will assess the evolution of the psychoneurological symptom cluster in two populations of patients with cancer: women with breast cancer, and patients with digestive cancer, over two years. Second, the investigators will test the feasibility and preliminary benefits of a new mind-body group intervention specifically designed to address the core symptom of the cluster, determined with network analysis in each population. As suggested by many authors, the proposed intervention will be based on the common-sense model of self-regulation developed by Leventhal and focus on cognitive-behavioral, self-care and mind-body (i.e., hypnosis) empowering strategies. The aim is to assess the satisfaction of the participants regarding the intervention, as well as its impact on the symptoms involved in the cluster.

ELIGIBILITY:
Inclusion critera for WP1:

* Diagnosis of non-metastatic breast cancer, or digestive cancer (i.e., anal, colorectal, gastric, esophageal, liver, pancreatic cancers).
* ≥ 18 years old.
* No history of cancer, and not currently in relapse.
* Having completed the active treatments (i.e., surgery, chemotherapy, radiotherapy) for 5 years maximum, based on the methodology and recommendations of studies on symptom clusters in oncology

Additional inclusion criteria for WP2:

* No history of severe psychiatric disorders (e.g., schizophrenia, dissociative episodes) or substance abuse (to avoid severe dissociation during hypnosis).
* Score ≥ 4 for the core symptom selected to design the intervention, as suggest by previous interventional studies, and measured on a visual analogue scale from 0 to 10.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2024-01-16 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Fatigue | WP1 : at inclusion (T0), then 6 months (T1), 12 months (T2) and 24 months (T3) later. WP2 : at inclusion (T0), then after the group sessions (T1, +- 2 months after T0).
  Assessed with a questionnaire (Multidimensional Fatigue Inventory; MFI-20). 5 subscales, each with a score comprised between 4 and 20, with a higher score indicating higher fatigue.
Change in pain | WP1 : at inclusion (T0), then 6 months (T1), 12 months (T2) and 24 months (T3) later. WP2 : at inclusion (T0), then after the group sessions (T1, +- 2 months after T0).
  Assessed with a visual analogue scale (VAS) (score range from 0 to 10/10, a higher score indicating a higher pain) and with a questionnaire (McGill Pain Questionnaire).
Change in sleep difficulties | WP1 : at inclusion (T0), then 6 months (T1), 12 months (T2) and 24 months (T3) later. WP2 : at inclusion (T0), then after the group sessions (T1, +- 2 months after T0).
  Assessed with a questionnaire (Insomnia Severity Index; ISI). Score range from 0 to 28, with a higher score indicating higher sleep difficulties.
Change in perceived cognitive difficulties | WP1 : at inclusion (T0), then 6 months (T1), 12 months (T2) and 24 months (T3) later. WP2 : at inclusion (T0), then after the group sessions (T1, +- 2 months after T0).
  Assessed with a questionnaire (FACT-Cog), investigation 4 dimensions (perceived cognitive impairments, score range 0-72, higher score indicating less impairments ; impact of cognitive impairments on quality of life, score range 0-16, with higher scoe indicating less impact ; Comments from others, score range 0-16 with higher score indicating less comments ; perceived cognitive abilities, score range 0-28, with higher score indicating more cognitive abilities)
Change in emotional distress | WP1 : at inclusion (T0), then 6 months (T1), 12 months (T2) and 24 months (T3) later. WP2 : at inclusion (T0), then after the group sessions (T1, +- 2 months after T0).
  Assessed with a questionnaire (Hospital Anxiety and Depression Scale; HADS). Score range from 0 to 42, with a higher score indicating higher emotional distress

SECONDARY OUTCOMES:
Change in quality of life | WP1 : at inclusion (T0), then 6 months (T1), 12 months (T2) and 24 months (T3) later. WP2 : at inclusion (T0), then after the group sessions (T1, +- 2 months after T0).
  Assessed with a core questionnaire (EORTC) and specific modules according to the cancer diagnosis (EORTC - ANL27, BR23, CR29, HCC18, OES18, OG25, PAN26, STO22). Score range varies according to the module. Higher score indicates a higher presence of the dimension investigated.
Change in self-compassion | WP1 : at inclusion (T0), then 6 months (T1), 12 months (T2) and 24 months (T3) later. WP2 : at inclusion (T0), then after the group sessions (T1, +- 2 months after T0).
  Assessed with a questionnaire (Self-compassion scale). Score range from 26 to 130, with higher score indicating higher self-compassion.
Change in self-care strategies | WP1 : at inclusion (T0), then 6 months (T1), 12 months (T2) and 24 months (T3) later. WP2 : at inclusion (T0), then after the group sessions (T1, +- 2 months after T0).
  Assessed with a questionnaire (self-care survey) consisting of a list of 24 strategies. For each of them, the participant indicates its frequency of use (occasionally, fairly often, very often) and its effectiveness to relieve fatigue (occasionally, fairly often, very often).
Change in coping strategies | WP1 : at inclusion (T0), then 6 months (T1), 12 months (T2) and 24 months (T3) later. WP2 : at inclusion (T0), then after the group sessions (T1, +- 2 months after T0).
  Assessed with a questionnaire (ways of coping checklist). Divided into 3 dimensions (i.e., problem-oriented coping, emotion-oriented coping, research of social support) with score ranging from 9 to 36. Higher score indicates a higher use of this kind of coping.
Change in perception about their fatigue | WP1 : at inclusion (T0), then 6 months (T1), 12 months (T2) and 24 months (T3) later. WP2 : at inclusion (T0), then after the group sessions (T1, +- 2 months after T0).
  Assessed with a questionnaire (Brief Illness Perception Questionnaire) composed of 8 VAS from 0 to 10.

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte GREGOIRE, PhD, Principal Investigator — University of Liege
Locations (1):
- University of Liège, Liège, Belgium

IPD SHARING:
Plan to Share IPD: Yes
The full protocol and anonymized data will be available upon reasonable request by email.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: When all data has been collected.
Access Criteria: by email (ch.gregoire@uliege.be)

REFERENCES:
- [Derived] Gregoire C, Baussard L, Ernst M, Diep A, Faymonville ME, Devos M, Jerusalem G, Vanhaudenhuyse A. Evaluation of a psychoneurological symptom cluster in patients with breast or digestive cancer: a longitudinal observational study. BMC Cancer. 2024 Jan 9;24(1):51. doi: 10.1186/s12885-023-11799-x. PMID 38195471